CLINICAL TRIAL: NCT02787265
Title: High-density in Spinal Cord Stimulation: Virtual Expert Registry
Acronym: Discover
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Moens Maarten, Prof. dr., Universitair Ziekenhuis Brussel
Other Study IDs: Discover1
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Failed Back Surgery Syndrome
Keywords: High density spinal cord stimulation; Virtual expert registry
MeSH Terms: conditions — Failed Back Surgery Syndrome | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (1):
- spinal cord stimulation: Failed back surgery syndrome patients will receive high density spinal cord stimulation
  Interventions: Device: spinal cord stimulation

INTERVENTIONS:
Device: spinal cord stimulation
  Other Names: high density spinal cord stimulation

SUMMARY:
This is a prospective, multi-center, observational follow-up study observing the effectiveness of high density spinal cord stimulation in patients with failed back surgery syndrome patients with back and leg pain.

DETAILED DESCRIPTION:
DISCOVER will measure the effectiveness of high-density spinal cord stimulation for treatment of chronic back and leg pain. Identification of clinical effective parameters concerning location of active electrodes, frequency, pulse duration, amplitude and battery consumption are, besides safety, the major outcome parameters of this study.

ELIGIBILITY:
Inclusion Criteria:

* Failed Back Surgery Syndrome patients (FBSS) with insufficient pain reduction with conventional SCS or FBSS patients suitable for SCS
* Age > 18 years
* Chronic pain as a result of FBSS that exists for at least 6 months with a pain intensity 5 or higher measured on numeric rating scale (NRS)
* Patient has been informed of the study procedures and has given written informed consent
* Patient willing to comply with study protocol including attending the study visits

Exclusion Criteria:

* Expected inability of patients to receive or properly operate the spinal cord stimulation system
* History of coagulation disorders, lupus erythematosus, diabetic neuropathy, rheumatoid arthritis or morbus Bechterew
* Active malignancy
* Addiction to any of the following drugs, alcohol (5E/day) and/or medication
* Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by investigator
* Immune deficiency (HIV positive, immunosuppressiva, etc.)
* Life expectancy < 1 year
* Local infection or other skin disorder at site of incision
* Pregnancy
* Other implanted active medical device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic back and leg pain (due to Failed Back Surgery Syndrome) who either received SCS or have not sufficient pain reduction with traditional parameters or patients with chronic back and leg pain who are candidate for SCS will receive HD SCS.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2016-06; Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity with the Numeric Rating Scale (NRS) | The difference between the baseline screening and the evaluation 1 month after high density stimulation, 3 months and 12 months.
Pain relief by pain medication | The difference between the baseline screening and the evaluation 1 month after high density stimulation, 3 months and 12 months.
  Questionnaire regarding the amount of pain relief by pain medication
The abilities in daily living | The difference between the baseline screening and the evaluation 1 month after high density stimulation, 3 months and 12 months.
  The functional abilities will be assessed with the Oswestry Low Back Pain Questionnaire.
The current health status | The difference between the baseline screening and the evaluation 1 month after high density stimulation, 3 months and 12 months.
  The health status will be observed with the Euroqol (EQ-5D-5L) questionnaire.
Subjective sleep quality | The difference between the baseline screening and the evaluation 1 month after high density stimulation, 3 months and 12 months.
  Subjective sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI).
Patient's satisfaction | The difference between the baseline screening and the evaluation 1 month after high density stimulation, 3 months and 12 months.
  Patient's satisfaction with the stimulation will be assessed with a 5 item Likert scale

SECONDARY OUTCOMES:
Pain area coverage | The difference between the evaluation 1 month after high density stimulation, 3 months and 12 months.
  The patient has to draw the areas of pain coverage on a body shape figure
Paresthesia threshold | The difference between the evaluation 1 month after high density stimulation, 3 months and 12 months.
  Patient indicates the threshold at which he experiences paresthesia
HD stim parameters | The difference between the evaluation 1 month after high density stimulation, 3 months and 12 months.
  Questionnaire towards the clinician regarding the ideal high density parameters for this patient
Battery efficiency of the neurostimulator | The difference between the evaluation 1 month after high density stimulation, 3 months and 12 months.
  The battery usage will be measured by frequencies to recharge the battery.
AdaptiveStim use (in case of Restore Sensor) | The difference between the evaluation 1 month after high density stimulation, 3 months and 12 months.
  Acquire information on activity from the internal diary; amount of times that patients need to fit the ideal parameters themselves
MRI need | The difference between the baseline screening and the evaluation 1 month after high density stimulation, 3 months and 12 months.
  Questionnaire regarding the need for MR scans for other medical conditions

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

REFERENCES:
- [Background] Song Z, Meyerson BA, Linderoth B. High-Frequency (1 kHz) Spinal Cord Stimulation-Is Pulse Shape Crucial for the Efficacy? A Pilot Study. Neuromodulation. 2015 Dec;18(8):714-20. doi: 10.1111/ner.12344. Epub 2015 Sep 6. PMID 26344573
- [Background] Sweet J, Badjatiya A, Tan D, Miller J. Paresthesia-Free High-Density Spinal Cord Stimulation for Postlaminectomy Syndrome in a Prescreened Population: A Prospective Case Series. Neuromodulation. 2016 Apr;19(3):260-7. doi: 10.1111/ner.12357. Epub 2015 Oct 20. PMID 26481726
- [Derived] Goudman L, Rigoard P, Billot M, De Smedt A, Roulaud M, Consortium D, Moens M; Discover Consortium. Spinal Cord Stimulation-Naive Patients vs Patients With Failed Previous Experiences With Standard Spinal Cord Stimulation: Two Distinct Entities or One Population? Neuromodulation. 2023 Jan;26(1):157-163. doi: 10.1016/j.neurom.2022.04.037. Epub 2022 May 10. PMID 35551868
- [Derived] Goudman L, De Smedt A, Eldabe S, Rigoard P, Linderoth B, De Jaeger M, Moens M; Discover Consortium. High-dose spinal cord stimulation for patients with failed back surgery syndrome: a multicenter effectiveness and prediction study. Pain. 2021 Feb 1;162(2):582-590. doi: 10.1097/j.pain.0000000000002035. PMID 32910099